CLINICAL TRIAL: NCT01980459
Title: Magnesium Treatment of Inflammation in Disorders of Glucose Homeostasis
Acronym: MagInGlu
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Nadia Zghoul, PhD, Dept of Clinical Research (Unknown); Dasman Diabetes Institute (Other)
Responsible Party: Principal Investigator, William Weglicki, Professor of Medicine, Biochemistry & Molecular Medicine, George Washington University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB#071317
Record Dates: First submitted 2013-10-22; First posted 2013-11-11 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Non-Insulin Dependent Diabetes Mellitus
Keywords: Hypomagnesemia, Cellular Mg, Inflammation, Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnesium Lactate (Experimental): Patients will receive 2 tablets twice a day of Magnesium Lactate for 3 months.
  Interventions: Dietary Supplement: magnesium lactate

INTERVENTIONS:
Dietary Supplement: magnesium lactate — Patient will be given 4 tablets a day of study supplement (Magnesium Lactate) for 3 months. Magnesium cellular and serum levels will be compared prior and post intervention.
  Other Names: MagTabSR

SUMMARY:
In most diabetic patients where low blood magnesium levels occur the important depletion of cellular levels is usually not measured. This study will measure both blood and oral mucosal cell magnesium levels before and after 3 months of supplementation with magnesium tablets (the recommended dietary amount of 336 milligrams per day). These magnesium levels will be correlated with blood levels of indicators of inflammation (eg C reactive protein) to see whether the cellular levels are more reliable than blood levels of magnesium for appropriate treatment of magnesium deficiency in diabetic patients.

DETAILED DESCRIPTION:
The anti-inflammatory effects of oral magnesium (Mg) supplementation of diabetic and metabolic syndrome patients with low serum Mg levels have been studied with increased interest in recent years. However, serum magnesium levels only represent less than one percent of total body magnesium; whereas cellular deficiency of Mg is a more reliable parameter to assess repletion of this essential mineral for correlation with indices of inflammation.

The proposed research will compare the efficacy of a 3 month period of treatment with oral Mg of diabetic patients selected for elevations of CRP, TNFα and other markers of inflammation on cellular and serum levels of Mg.

We anticipate that 50 hypomagnesemic diabetic patients will be selected for 3 months of supplementation with 336 mg of Mg lactate tablets. The repletion of serum and oral epithelial cell Mg levels will be correlated with responses of CRP, TNFα, substance P, HgbAIc and oxidative/nitrosative (ROS/RNS) stress parameters before and after treatment. Individuals will be selected from the Dasman Diabetes Institute in Kuwait. With completion of these analyses, a collaborative manuscript with joint authorship will be prepared and submitted for publication.

ELIGIBILITY:
Inclusion Criteria:

* Have documented hypomagnesemia (serum levels ≤ 1.8 mg/dL or 0.74mmol/L);
* Be between 20-70 years of age at the time of randomization
* Have hyperglycemia due to NIDDM metabolic syndrome or obesity
* Have at least one abnormal indicator of inflammation (e.g. elevated CRP, TNF-α)
* Have no active infection

Exclusion Criteria:

* Currently have significant gastrointestinal disorders (e.g. chronic diarrhea);
* Have impaired renal function, defined as eGFR < 60 mL/min/1.73m2 or serum creatinine > 1.3 mg/dL;
* Are current being treated for hypertension (e.g. ACE inhibitors and diuretics), heart block (e.g. EKG evidence of left bundle branch block) or heart failure (e.g. treated with aldosterone antagonists);
* Are currently pregnant;
* Have chronic inflammatory disorders (e.g. psoriasis);
* Have used of Mg supplements and Mg-rich mineral water within 6 months;

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The magnesium cellular levels will provide a stronger correlation with antiinflammatory indicators compared to the circulating serum levels of magnesium. | One year
  50 hypomagnesemic diabetic patients will receive magnesium tablets (~recommended dietary allowance)for 3 months and circulating inflammatory indicators will be measured. The blood and cellular levels of magnesium will be measured (before and after treatment) to assess which parameter correlates best with efficacy in lowering inflammation indicators.

SECONDARY OUTCOMES:
Magnesium supplementation will lower parameters of inflammation in hypomagnesemic diabetic patients. | One year
  Antiinflammatory indicators (CRP, TNF alpha, isoprostane, Hemoglobin A1c etc) will be measured prior to and after 3 months of magnesium supplementation .

CONTACTS AND LOCATIONS:
Overall Officials: William B Weglicki, MD, Principal Investigator — George Washington University; Nadia Zghoul, PhD, Principal Investigator — Dasmin Diabetes Institute
Locations (1):
- The Dasman Diabetes Institute, Kuwait City, Kuwait